CLINICAL TRIAL: NCT06674941
Title: A Phase 1, Open-label, Single-dose Trial to Evaluate the Pharmacokinetics, Safety and Tolerability of Teprotumumab (High-concentration Formulation) Subcutaneous Administration in Healthy Adult Non-Japanese and Japanese Volunteers
Brief Title: A Trial to Investigate Teprotumumab (High-concentration Formulation) Subcutaneous Administration in Healthy Adult Non-Japanese and Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HZNP-TEP-104
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Healthy Volunteers
Keywords: Thyroid eye disease; Graves' ophthalmopathy; Graves' orbitopathy; Thyroid-associated ophthalmopathy; Immunology
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — teprotumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: Teprotumumab (Experimental): Non-Japanese participants will receive SC injection of teprotumumab Dose A by a syringe pump.
  Interventions: Drug: Teprotumumab
- Cohort 2: Teprotumumab (Experimental): Japanese participants will receive SC injection of teprotumumab Dose A by a syringe pump.
  Interventions: Drug: Teprotumumab
- Cohort 3: Teprotumumab (Experimental): Non-Japanese participants will receive SC injection of teprotumumab Dose B by an injection device.
  Interventions: Drug: Teprotumumab

INTERVENTIONS:
Drug: Teprotumumab — Administered as an SC injection.
  Other Names: Teprotumumab-trbw; TEPEZZA; HZN-001

SUMMARY:
The primary objective of this trial are to assess the pharmacokinetics (PK) of a single subcutaneous (SC) administration of teprotumumab high-concentration formula (HCF) in healthy adult non-Japanese and Japanese participants and to assess the PK of teprotumumab delivered by syringe pump and by an injection device in non-Japanese participants.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is a healthy male or female between the ages of 18 and 55 years, inclusive, at Screening.
2. Participant has a body mass index between 18 and 30 kg/m^2, inclusive, at Screening.
3. Participant is medically healthy, with no clinically significant medical history, physical examination, laboratory profiles, vital signs, or 12-lead ECG results at Screening, as deemed by the Principal Investigator (PI) or designee.
4. If female of childbearing potential (including those with an onset of menopause < 2 years prior to Screening, non-therapy-induced amenorrhea for < 12 months prior to Screening or not surgically sterile [absence of ovaries and/or uterus]) must have a negative serum pregnancy test at Screening and Check-in and negative urine pregnancy tests at all protocol-specified time points (ie, prior to the teprotumumab dose and throughout participation in the Follow-up Period); female participants of childbearing potential who are sexually active with a non-vasectomized male partner must agree to use 2 reliable forms of contraception during the trial, 1 of which is recommended to be hormonal, such as an oral contraceptive. Hormonal contraception must be started at least 1 full cycle prior to Day 1 and continue for 180 days after receiving the dose of teprotumumab. Highly effective contraceptive methods (with a failure rate < 1% per year), when used consistently and correctly, include implants, injectables, combined oral contraceptives, some intrauterine devices, vasectomized partner, or sexual abstinence. Abstinence should only be used as a contraceptive method if it is in line with the participant usual and preferred lifestyle. Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods) is not an acceptable method of contraception.
5. If female, participant must agree not to donate an egg/oocyte from Day 1 until 180 days after receiving the dose of teprotumumab.
6. If male, participant must be surgically sterile for at least 6 months prior to dosing or, if sexually active with a female partner of childbearing potential, must agree to use a barrier contraceptive method from Screening through 180 days after receiving the dose of teprotumumab.
7. If male, must agree not to donate sperm from Day 1 until 180 days after receiving the dose of teprotumumab.
8. Participant has adequate venous access.
9. Participant understands the trial procedures in the ICF and is willing and able to comply with the prescribed treatment protocol and evaluations for the duration of the trial.

   Additional Inclusion Criteria for Cohort 2:
10. First generation Japanese healthy male or female participants must meet all of the following as confirmed by interview:

    1. Descendants of 4 ethnic Japanese grandparents who were born in Japan
    2. Both parents are ethnic Japanese who were born in Japan
    3. Hold a Japanese passport or identity papers
    4. Have lived outside Japan for less than 10 years at the time of screening and lifestyle including diet has not changed significantly since leaving Japan.

Exclusion Criteria:

1. Participant has a history or presence of a clinically significant medical or psychiatric condition or disease, in the opinion of the PI or designee.
2. Participant has a history of any illness that, in the opinion of the PI or designee, might confound the results of the trial or pose an additional risk to the participant due to participation in the trial.
3. Participant has a history or presence of alcoholism (defined as > 10 standard drinks per week, where 1 standard drink = 284 mL of full-strength [4.9% alc/vol] beer, 30 mL of 40% [alc/vol] spirit or a 100 mL glass of wine]) or drug abuse within the 6 months prior to Day 1 dosing.
4. Participant has a history or presence of hypersensitivity or idiosyncratic reaction to components of teprotumumab or prior hypersensitivity reactions to a monoclonal antibody or history.
5. Participant has a history or presence of:

   1. thyroid eye disease
   2. diagnosis of autoimmune diseases
   3. inflammatory bowel disease
6. Participant has an alanine transaminase or aspartate transaminase level > 1.5 times upper limit of normal at Screening or Check-in.
7. Participant has glycated hemoglobin ≥ 6.5% and/or fasting glucose level (after at least an 8-hour fast) > 126 mg/dL at Screening.
8. Participant has clinically significant abnormal ECG measurements at Screening or prior to teprotumumab dosing, in the opinion of the PI, or has second- or third-degree atrioventricular block or any of the following:

   1. QRS > 120 msec
   2. QTcF) > 450 msec (males) or > 470 msec (females)
   3. PR interval > 220 msec
9. Participant has a medical condition associated with increased risk of bleeding, including history of hematological diseases such as acquired platelet disorders and coagulation disorders, including drug-induced thrombocytopenia, idiopathic thrombocytopenia or von t medication.
10. Participant has donated blood, has had significant blood loss, or has received a transfusion of any blood or blood products within 60 days prior to Day 1 or plasma donation within 7 days prior to Day 1.
11. Participant has participated in another clinical trial within 30 days (or 5 half-lives of the trial drug, whichever is longer) prior to Day 1. The 30-day (or 5 half-lives) window will be derived from the date of last dosing in the previous trial to the date of Day 1 of the current trial.
12. Participant has previous participation in a teprotumumab clinical trial or received teprotumumab or any anti-human insulin-like growth factor-1 receptor monoclonal antibody.
13. Participant has any other condition that, in the opinion of the Investigator, would preclude inclusion in the trial.
14. Participant has used any prescription (excluding hormonal birth control) or over-the-counter medications, including herbal or nutritional supplements, within 14 days before receiving the study drug. Over-the-counter use of acetaminophen (up to 2 g per day), topical eye drops, and topical creams are allowed. Use of other over-the-counter medications may be allowed at the discretion of Investigator with approval from the Medical Monitor.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2023-03-24 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-14 (Actual)

PRIMARY OUTCOMES:
Area Under the Serum Concentration-time Curve (AUC) From Time 0 Extrapolated to Infinity (AUCinf) of Teprotumumab | Day 1 pre-dose to Day 57
AUC From Time 0 to the Last Quantifiable Concentration (AUClast) of Teprotumumab | Day 1 pre-dose to Day 57
Maximum Observed Serum Concentration (Cmax) of Teprotumumab | Day 1 pre-dose to Day 57
Time to Cmax (Tmax) of Teprotumumab | Day 1 pre-dose to Day 57

SECONDARY OUTCOMES:
Number of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | Up to Day 57
  Number of participants with TEAEs, severe TEAEs, infusion-related reactions, injection-site reactions, and adverse device effects will be reported. Clinically significant changes in laboratory tests, vital signs and electrocardiograms (ECG) will be reported as adverse events.
Number of Participants with Anti-drug Antibodies (ADA) to Teprotumumab | Day 1 pre-dose to Day 57
Titer of Positive ADA to Teprotumumab | Day 1 pre-dose to Day 57

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- PPD Development, LP, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com